CLINICAL TRIAL: NCT00722059
Title: Assessment of Emerging Technology: Comparison of Breast Tomosynthesis and Digital Mammography in the Evaluation of Heterogeneously Dense and Extremely Dense Breasts
Brief Title: Detection and/or Evaluation of Dense Breast Abnormalities Using Tomosynthesis and Digital Mammography
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Alexis V. Nees M.D., Principal Investigator, University of Michigan
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HUM 13236
Record Dates: First submitted 2008-07-23; First posted 2008-07-25 (Estimated); Last update posted 2014-02-03 (Estimated); Status verified 2014-01

CONDITIONS: Breast Neoplasms; Breast Abnormalities
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Subjects will undergo a 3D breast Tomosynthesis imaging scan. This is a one time breast imaging scan will last approximately 15 minutes.
  Interventions: Procedure: Breast Tomosynthesis

INTERVENTIONS:
Procedure: Breast Tomosynthesis — 3D breast imaging

SUMMARY:
The purpose of this study is to compare 3D mammography with digital mammography in women with dense breasts for the detection and evaluation of masses and/or breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Females 30 years of age or older.
* Dense Breasts.
* Has undergone clinical two view mammogram and diagnostic breast imaging evaluation.
* Suspicious or palpable mass and scheduled for biopsy.

Exclusion Criteria:

* Pregnant or lactating women.
* Prior personal history of breast cancer.
* Prior breast augmentation with implants or silicon injection. male patients.
* No two view mammogram as part of breast imaging evaluation.
* Breast density of almost entirely fatty/scattered fibroglandular densities.

Min Age: 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2006-04; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Measure of digital tomosynthesis and digital mammography test performance. | 3 weeks
  Interest of sensitivity, specificity and area under region of concern curve for malignant mass detection. During review, the number of masses and location and size of each mass will be recorded. An additional estimate of probability of malignancy will be recorded for each image sets.

CONTACTS AND LOCATIONS:
Overall Officials: Alexis V. Nees, M.D., Principal Investigator — University of Michigan
Locations (1):
- University of Michigan Health System, Ann Arbor, Michigan, United States